CLINICAL TRIAL: NCT02023619
Title: Comparison of Corneal Epithelial and Stromal Thickness Distributions Between Eyes With Keratoconus and Healthy Eyes With Corneal Astigmatism >2.0 D
Brief Title: Corneal Epithelial and Stromal Thickness Distribution in Keratoconus
Status: Completed | Type: Observational
Sponsor: SynsLaser Kirurgi AS (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Aleksandar Stojanovic, Medical director of SynsLaser Surgery AS, SynsLaser Kirurgi AS
Other Study IDs: REK NORD 2013/758; SL 1 (Other: SynsLaser)
Record Dates: First submitted 2013-12-12; First posted 2013-12-30 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Keratoconus; Astigmatism
Keywords: Keratoconus; Astigmatism; Cornea; SD-OCT
MeSH Terms: conditions — Keratoconus; Astigmatism; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Keratoconus: Eyes with confirmed keratoconus diagnosis
- Astigmatism >2.0 D: Healthy eyes with astigmatism >2.0 D

SUMMARY:
The purpose of the study was to identify corneal epithelial- and stromal-thickness distribution patterns in keratoconic eyes using spectral-domain-optical coherence tomography (SD-OCT).

Study Hypothesis: SD-OCT provides necessary details about the distribution of corneal epithelial and stromal thicknesses for identification of a pattern characteristic for early keratoconus.

DETAILED DESCRIPTION:
Purpose of the study: To characterize epithelial and stromal thickness distribution in keratoconic eyes and to develop epithelial and stromal thickness-based variables for keratoconus detection.

Methodology: SD-OCT corneal scans of 20 eyes with keratoconus (group 1) and 20 healthy eyes with > 2 diopters (D) of corneal astigmatism as controls (group 2) are studied. Keratoconus patients referred to the Eye Dpt. of the University Hospital North Norway for CXL (Corneal collagen cross-linking)- treatment and healthy subjects seeking preoperative evaluation for refractive surgery at SynsLaser® Kirurgi AS Tromsø clinic are examined by corneal SD-OCT as a part of their routine examination. Analysis of their SD-OCT corneal scans is used for the purpose of this study.Two cross-sectional meridional corneal profiles (along steepest and flattest meridians, located by a Scheimpflug-based corneal topography) for each individual are obtained by using a RTVue100® (Optovue Inc. Fremont, California, USA), 26000-Hz SD-OCT across the central 6mm diameter of the cornea.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus group: Confirmed diagnosis of keratoconus
* Astigmatism group: Healthy eyes with astigmatism of >2.0 D

Exclusion Criteria:

* Keratoconus group: Keratoconus > stage 3 on Krumeich scale
* Astigmatism group: No signs of keratoconus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 eyes with diagnosed keratoconus and 20 healthy eyes with astigmatism >2.0 D
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cornea epithelial thickness distribution | Up to 24 weeks
  A single non-invasive measurement by OCT evaluated up to 24 weeks after the examination

SECONDARY OUTCOMES:
Cornea stromal thickness distribution | Up to 24 weeks
  A single non-invasive measurement by OCT evaluated up to 24 weeks after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Stojanovic, MD, Principal Investigator — SynsLaser Kirurgi AS
Locations (1):
- SynsLaser Kirurgi AS, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou W, Stojanovic A. Comparison of corneal epithelial and stromal thickness distributions between eyes with keratoconus and healthy eyes with corneal astigmatism >/= 2.0 D. PLoS One. 2014 Jan 28;9(1):e85994. doi: 10.1371/journal.pone.0085994. eCollection 2014. PMID 24489687